CLINICAL TRIAL: NCT03761030
Title: Targeting Dopaminergic Mechanisms of Slowing to Improve Late Life Depression
Brief Title: L-DOPA vs. Placebo for Depression and Psychomotor Slowing in Older Adults
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The project end date was reached prior to the full sample enrollment
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bret Rutherford, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7733; 4R33MH110029-03 (NIH)
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Major Depressive Disorder; Dysthymia; Depression
Keywords: Depressive symptoms; Cognitive problems; Antidepressant non-response; Dopamine system; Older Adults; Motor slowing
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Depression | interventions — Levodopa; Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-DOPA Arm (Experimental): Those assigned to L-DOPA will begin taking 37.5mg carbidopa/150 mg levodopa once daily (with placebo twice daily) for one week, then increase to 75mg carbidopa/300mg levodopa (37.5 mg carbidopa/150mg levodopa twice daily and placebo once daily) for one week, and finally increase to 112.5mg carbidopa/450mg levodopa (37.5 mg carbidopa/150mg levodopa three times daily and no placebo) for the final six weeks. Each subject assigned to the L-DOPA arm will be titrated to 450mg L-DOPA unless they cannot tolerate higher doses, in which case subjects will have their dosage reduced to the maximum tolerable dose
  Interventions: Drug: L-DOPA
- Placebo Arm (Placebo Comparator): Subjects assigned to the placebo arm will take placebo oral tablet three times daily throughout the study.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: L-DOPA — We will be using generic sinemet 25/100 tablets in this study.
  Other Names: carbidopa/levodopa (Sinemet)
  Arms: L-DOPA Arm
Drug: Placebo Oral Tablet — 25/100 placebo tablets
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
Individuals with Late Life Depression (LLD) often have cognitive problems, particularly problems with memory, attention, and problem solving, all of which contribute to antidepressant non-response. Our group and others have shown that decreased thinking speed is the central cause of functional problems in patients with LLD. Similarly, decreased walking speed is associated with depression and carries additional risk for falls, hospitalization, and death. Available evidence suggests that declining functionality in the brain's dopamine system contributes to age-related cognitive and motor slowing. The central hypothesis of this study is that by enhancing dopamine functioning in the brain and improving cognitive and motor slowing, administration of carbidopa/levodopa (L-DOPA) will improve depressive symptoms in older adults.

DETAILED DESCRIPTION:
Enrolled participants were aged 60 and older with (1) a DSM 5 depressive disorder, (2) significant depressive symptoms, and (3) decreased thinking or walking speed will receive 8 weeks of treatment with L-DOPA up to 450mg. We will test whether L-DOPA increases brain dopamine release using neuroimaging and whether it speeds up thinking and walking speed. Data collected in the proposed studies may help identify a new treatment for LLD, which could have large public health ramifications given the prevalence, frequent treatment resistance, and chronicity characteristic of LLD. This project also will elucidate the neurobiology of slowing at molecular, structural, and functional levels of analysis, increasing our understanding of the interplay between these aging-associated processes and the pathophysiologic changes underlying late life neuropsychiatric disorders. Exploring patient characteristics that predict response to L-DOPA may provide useful information to guide differential therapeutics and develop personalized medicine for LLD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 years and older
2. DSM 5 non-psychotic Major Depressive Disorder, Dysthymia, or Depression Not Otherwise Specified
3. Hamilton Rating Scale for Depression (HRSD) > 15
4. Decreased processing speed (defined as performance > 0.5SD below age-adjusted norms on Digit Symbol Substitution Test or Trail Making Test Part A) OR decreased gait speed (defined as average walking speed over 15' course < 1m/s)
5. Willing to and capable of providing informed consent and complying with study procedures
6. Alternative standard treatments for MDD, Dysthymia, or Depression NOS (e.g., antidepressant medication or psychotherapy) have been discussed and the individual agrees to be involved in an experimental treatment.

Exclusion Criteria:

1. Diagnosis of substance abuse or dependence (excluding Tobacco Use Disorder) within the past 12 months.
2. History of or current psychosis, psychotic disorder, mania, or bipolar disorder
3. Diagnosis of probable Alzheimer's Disease, Vascular Dementia, or Parkinson's Disease (PD)
4. Mini Mental Status Exam (MMSE) < 25
5. HRSD ≥ 28; HRSD suicide item > 2 or the presence of significant suicide risk as judged by clinician or Clinical Global Impressions (CGI)-Severity score of 7 at baseline.
6. Current or recent (within the past 4 weeks) treatment with antidepressants, antipsychotics, dopaminergic agents, or mood stabilizers.
7. History of allergy, hypersensitivity reaction, or severe intolerance to L-DOPA
8. Acute, severe, or unstable medical or neurological illness
9. Mobility limiting osteoarthritis of any lower extremity joints, symptomatic lumbar spine disease, mobility limiting history of joint replacement surgery, or history of spine surgery

   FOR SUBJECTS RECEIVING PET/MRI SCANS ONLY:
10. Having contraindication to MRI scanning (such as metal in body) or unable to tolerate the scanning procedures
11. History of significant radioactivity exposure (nuclear medicine studies or occupational exposure)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 51 subjects were enrolled. Of the 51 enrolled, 20 subjects were found to be ineligible or did not continue in the study after enrolling. Thus, 51 participants enrolled and 31 were assigned to a treatment group and began the study.
Period: Overall Study
Arm/Group | L-DOPA Arm | Placebo Arm
Started | 15 | 16
Completed | 13 | 12
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-DOPA Arm | Placebo Arm | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (7.3) | 66.7 (6.1) | 67.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 9 | 10 | 19
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31
Hamilton Rating Scale for Depression (24 item) [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Rating Scale for Depression (HRSD) is a 24-item questionnaire used as an indication of depression and a guide to evaluate recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score of 16 or above is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity.
  units on a scale | 21.1 (4.7) | 20.3 (3.9) | 20.7 (4.3)
Clinical Global Impressions--Severity [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impressions--Severity (CGI-S) scale measures the clinician's assessment of global illness severity. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Higher scores denote more severe illness.
  units on a scale | 3.7 (0.6) | 4.3 (0.7) | 4.0 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Hamilton Rating Scale for Depression 24-Item Scale to Study Completion (8 Weeks)
Description: The Hamilton Rating Scale for Depression (HRSD) is a 24-item questionnaire used as an indication of depression and a guide to evaluate recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score of 16 or above is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 8 Weeks
Population: Participants with Week 8 data available were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | L-DOPA Arm | Placebo Arm
Number analyzed (Participants) | 12 | 13
units on a scale | -2.2 (6.4) | -3.6 (5.8)

2. Secondary Outcome: Digit Symbol Test
Description: The Digit Symbol test is a neuropsychological test measuring information processing speed. It consists of digit-symbol pairs (e.g. 1/-,2/┴ ... 7/Λ,8/X,9/=) followed by a list of digits. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time is measured. Score ranges from 0-133, with higher scores indicating higher information processing speed. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 8 Weeks
Population: Participants with Week 8 data available were analyzed.
Measure: Mean (Standard Deviation); unit: Number of items correctly completed
Arm/Group | L-DOPA Arm | Placebo Arm
Number analyzed (Participants) | 9 | 10
Number of items correctly completed | 2.8 (4.0) | 5.0 (3.5)

3. Secondary Outcome: Single Task Gait Speed
Description: Patients' gait was assessed as walking speed in cm/s on a 15' walking course. Patients walked at their usual or normal speed for a total of 27' (starting and ending at a point 6 feet prior to and after the 15' course to eliminate acceleration and deceleration effects). Two trials were completed, and gait speed was based on the average of 2 trials. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 8 Weeks
Population: Participants with Week 8 data available were analyzed
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | L-DOPA Arm | Placebo Arm
Number analyzed (Participants) | 10 | 9
cm/s | 3.7 (14.9) | -3.8 (14.7)

4. Secondary Outcome: Inventory of Depressive Symptomatology--Self Report (IDS-SR)
Description: The Inventory of Depressive Symptomatology--Self Report (IDS-SR) is a rating scale for depressive symptoms based on standard diagnostic criteria for Major Depressive Disorder. The scale ranges from 0-84 with higher scores indicating more severe depression. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 8 Weeks
Population: Participants with available Week 8 data were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | L-DOPA Arm | Placebo Arm
Number analyzed (Participants) | 10 | 10
units on a scale | -9.8 (7.1) | -12.1 (15.0)

5. Secondary Outcome: Pattern Comparison Test
Description: This test required participants to identify whether two visual patterns are the "same" or "not the same" (responses were made by pressing a "yes" or "no" button). Patterns were either identical or varied on one of three dimensions: color (all ages), adding/taking something away (all ages), or one versus many. Scores reflect the number of correct items completed in 90 s, with scores ranging from a minimum of 0 to a maximum of 30. Items were designed to minimize the number of errors that were made. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 8 Weeks
Population: Participants with available Week 8 data were analyzed
Measure: Mean (Standard Deviation); unit: Number of items correctly completed
Arm/Group | L-DOPA Arm | Placebo Arm
Number analyzed (Participants) | 11 | 10
Number of items correctly completed | 0.6 (2.1) | 1.2 (2.3)

6. Secondary Outcome: Letter Comparison Test
Description: Subjects were asked to determine whether two strings of letters are the same or different. There are 3 pages and the subject is given 30 seconds per page. Scoring is based on the number answered correctly. Scores range from 0 to 21, with the higher the number, the better the score. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 8 Weeks
Population: Participants with available Week 8 data were analyzed
Measure: Mean (Standard Deviation); unit: Number of items correctly completed
Arm/Group | L-DOPA Arm | Placebo Arm
Number analyzed (Participants) | 11 | 10
Number of items correctly completed | 1.2 (1.6) | 0.7 (1.4)

ADVERSE EVENTS:
Time Frame: Subjects were monitored over a period of 8 weeks.
Arm/Group | L-DOPA Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/16
Other Adverse Events (participants affected / at risk) | 14/15 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-DOPA Arm (N=15) | Placebo Arm (N=16)
Hospitalization for infection (Infections and infestations) | 0 (0) | 1 (1)
Death by suicide (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-DOPA Arm (N=15) | Placebo Arm (N=16)
Blurred vision (Eye disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (8) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3)
Stomach/throat discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Increased appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hot flashes (General disorders) | 2 (2) | 0 (0)
Malaise/weakness (General disorders) | 1 (1) | 2 (2)
Poor balance (General disorders) | 1 (1) | 1 (1)
Incidental MRI finding (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety during neuroimaging (Psychiatric disorders) | 0 (0) | 2 (2)
Fall (General disorders) | 0 (0) | 1 (1)
Toe fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck/back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
Joint/limb pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Leg/ankle swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle tightness/rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Numbness (Nervous system disorders) | 1 (1) | 0 (0)
Word finding difficulty (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (7) | 6 (7)
Drowsiness (Psychiatric disorders) | 5 (6) | 2 (2)
Excitement (Psychiatric disorders) | 2 (2) | 0 (0)
Vivid dreams (Psychiatric disorders) | 1 (1) | 3 (3)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Forgetfulness (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Panic (Psychiatric disorders) | 0 (0) | 1 (1)
Increased urination (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Cloudy urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Sighing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Increased sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dizziness (Vascular disorders) | 6 (6) | 4 (4)
Increased heart rate (Vascular disorders) | 2 (2) | 0 (0)
Decreased heart rate (Vascular disorders) | 1 (1) | 1 (1)
Abnormal heart rhythm (Vascular disorders) | 1 (1) | 0 (0)
Palpitations (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Data collected in the trial have been presented as required but are considered unreliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT03761030/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03761030/SAP_001.pdf
  • Informed Consent Form (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT03761030/ICF_002.pdf